CLINICAL TRIAL: NCT04460001
Title: Intravitreal Injection of Ranibizumab Versus Combination of Ranibizumab and Triamcinolone Acetate for the Treatment of Macular Edema Secondary to Central Retinal Vein Occlusion (CRVO)
Brief Title: Injection of Ranibizumab Versus Combination of Ranibizumab and Triamcinolone Acetate for (CRVO)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Wael Ali Mohamed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WAMohamed
Record Dates: First submitted 2019-08-01; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2019-11

CONDITIONS: Ophthalmopathy
MeSH Terms: conditions — Eye Diseases | interventions — Ranibizumab; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranibizumab (Active Comparator): intravetreal injection of Ranibizumab alone for treatment of patients with macular oedema after CRVO once per month and follow up
  Interventions: Drug: Ranibizumab
- Ranibizumab and triamcinolone acetate (Active Comparator): intravetreal injection of Ranibizumab and triamcinolone acetate for treatment of patients with macular oedema after CRVO once per month and follow up
  Interventions: Drug: Ranibizumab; Drug: triamcinolone acetate

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal
  Arms: Ranibizumab
Drug: Ranibizumab — Intravitreal
  Arms: Ranibizumab and triamcinolone acetate
Drug: triamcinolone acetate — intravitreal
  Arms: Ranibizumab and triamcinolone acetate

SUMMARY:
To compare the clinical effectiveness of ranibizumab and combination of ranibizumab and triamcinolone for the treatment of macular oedema secondary to CRVO

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with visual impairment resulting from macular edema secondary to CRVO.
* A BCVA approximate Snellen equivalents, 20/40.

Exclusion Criteria:

* Use of intra-vitreal anti-VEGF injections 3 months or less before baseline.
* Pan-retinal laser photocoagulation 3 months or less before baseline,
* Topical ocular or systemic corticosteroids administered for 30 consecutive days.
* Intraocular or periocular corticosteroid use 3 months or less before screening (study eye),
* Use of intraocular corticosteroid implants,
* Uncontrolled glaucoma (intraocular pressure [IOP] 30 mmHg with medication) at the time of screening or baseline,
* iris neovascularization or neo-vascular glaucoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between intravitreal injection of ranibizumab and combination of ranibizumab and triamcinolone acetate for the treatment of macular edema secondary to CRVO | 2 year
  To compare the clinical effectiveness of 0.5 mg ranibizumab and combination of ranibizumab and triamcinolone 0.3/0.5mg for the treatment of macular oedema secondary to CRVO.Study assessments will be performed at screening, baseline and at monthly visits:
  Best-Corrected Visual Acuity:
  will be assessed at every study visit by using alandolt ringes VA testing chart at an initial testing distance of 6 m.
Comparison between intravitreal injection of ranibizumab and combination of ranibizumab and triamcinolone acetate for the treatment of macular edema secondary to CRVO | 2 year
  To compare the clinical effectiveness of 0.5 mg ranibizumab and combination of ranibizumab and triamcinolone 0.3/0.5mg for the treatment of macular oedema secondary to CRVO.Study assessments will be performed at screening, baseline and at monthly visits:
  Optical Coherence Tomography:
  will be performed at every visit and the same machine will be used for assessment of the same patient throughout the study. investigator will evaluate the images according to central foveal thickness, and the retinal thickness at the foveal center point and to capture the presence or absence of qualitative parameters (i.e., intraretinal cystoid fluid and subretinal fluid).

CONTACTS AND LOCATIONS:
Locations (1):
- Wael, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided